CLINICAL TRIAL: NCT05959616
Title: Safety and Feasibility of a Shigella Sonnei 53G Controlled Human Infection Model in Kenyan Adults: a Dose Finding and Dose Verification Study
Brief Title: Shigella Sonnei 53G Human Infection Study in Kenyan Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: KEMRI-Wellcome Trust Collaborative Research Program (Other); KEMRI United States Army Medical Research Directorate-Kenya (Unknown); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Naval Medical Research Center (U.S. Federal Agency); PATH (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: OxTREC27-22
Record Dates: First submitted 2023-06-29; First posted 2023-07-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-05

CONDITIONS: Shigellosis
MeSH Terms: conditions — Dysentery, Bacillary | interventions — Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Group 1 Shigella sonnei 53G 1500CFU (N=10) (Experimental): Dose finding group
  Group 1 will receive lyophilised S. sonnei 53G strain at a dose of 1500CFU.
  Group 1 will receive curative treatment of Ciprofloxacin.
  Interventions: Biological: Shigella sonnei 53G; Drug: Ciprofloxacin 500 mg
- Group 2 Shigella sonnei 53G 2000CFU (N=10) (Experimental): Dose finding group
  Group 2 will receive lyophilised S. sonnei 53G strain at a dose of 2000CFU.
  Group 2 will receive curative treatment of Ciprofloxacin.
  Interventions: Biological: Shigella sonnei 53G; Drug: Ciprofloxacin 500 mg
- Group 3 Shigella sonnei 53G 2500CFU (N=10) (Experimental): Dose finding group
  Group 3 will receive lyophilised S. sonnei 53G strain at a dose of 2500CFU.
  Group 3 will receive curative treatment of Ciprofloxacin.
  Interventions: Biological: Shigella sonnei 53G; Drug: Ciprofloxacin 500 mg
- Group 4 Shigella sonnei 53G 3000CFU (N=10) (Experimental): Dose finding group
  Group 4 will receive lyophilised S. sonnei 53G strain at a dose of 3000CFU.
  Group 4 will receive curative treatment of Ciprofloxacin.
  Interventions: Biological: Shigella sonnei 53G; Drug: Ciprofloxacin 500 mg
- Group 5 Shigella sonnei 53G TBDCFU (N=15) (Experimental): Dose verification group
  Group 5 will receive lyophilised S. sonnei 53G strain at a dose TBD.
  Group 5 will receive curative treatment of Ciprofloxacin.
  Interventions: Biological: Shigella sonnei 53G; Drug: Ciprofloxacin 500 mg
- Group 6 Shigella sonnei 53G TBDCFU (N=15) (Experimental): Dose verification group
  Group 6 will receive lyophilised S. sonnei 53G strain at a dose TBD.
  Group 6 will receive curative treatment of Ciprofloxacin.
  Interventions: Biological: Shigella sonnei 53G; Drug: Ciprofloxacin 500 mg

INTERVENTIONS:
Biological: Shigella sonnei 53G — Lyophilized S. sonnei 53G strain (Lot 1794)
Drug: Ciprofloxacin 500 mg — Ciprofloxacin (500 mg orally twice daily for three days),

SUMMARY:
Diarrhoea caused by Shigella (shigellosis) is of major public health importance. However, there are no licensed Shigella vaccines in routine use, with several candidates still in various stages of clinical development. Shigella human infection studies (HIS) have played a key role in vaccine development. These models also allow for the evaluation of immunity and other non-immunological parameters that are important to understand resistance and/or susceptibility to disease. This is particularly useful in individuals from endemic areas with varying levels of prior exposure and immunity to Shigella. Thus, establishing a Shigella HIS would enable the testing of interventions such as vaccines in a population that would most benefit from a subsequent vaccine and has potential to accelerate vaccine development. Here, the goal is to successfully establish a Shigella sonnei human infection model in Kenyan adults. This will be achieved by conducting dose-finding and dose verification Shigella studies that safely and reproducibly induce ≥60% attack rates. In this study, investigators aim to use Shigella HIS in healthy adults to develop a model as a platform to test vaccines, to study immune responses identifying potential correlates of infection, and non-immunological factors mediating and influencing susceptibility to disease. To achieve this, the study will be carried out in two phases over a period of 12-14 months. Phase A will enroll (N=up to 40 volunteers) and Phase B will enroll an additional (N=30 volunteers). To be eligible to receive a dose of 53G, volunteers must pass the screening visit. Investigators will vary the dose of bacteria in individuals enrolled for challenge to identify the dose needed to cause ≥60% shigellosis (attack rate) (Phase A) followed by testing and demonstrate the reproducibility of the model (Phase B). Thus, the main outcomes of the study will be: (1) optimisation of bacterial dose for infection success (≥60% attack rate); and (2) safety.

DETAILED DESCRIPTION:
This is a Phase 1 dose finding and dose verification study which will be used to determine the dose of S. sonnei 53G that induces the primary outcome in approximately ≥60% of Kenyan adult volunteers. This study will occur in two phases, Phase A (dose-finding) with up to 40 volunteers challenged with 53G and Phase B (dose verification) with N=30 volunteers planned to be administered 53G. Based on previously published data using this model, 1,500 colony-forming units (CFU) will be the dose administered to the first cohort. Dosing of subsequent cohorts will depend on results of the previous cohort. If a lower-than-expected attack rate (AR) occurs, the dose for the next cohort will be increased by 500 CFU. Conversely, if the AR is higher than expected the dose for the next cohort will be decreased by 500 CFU. Cohorts of volunteers will continue to be challenged until either; a dose that reproducibly causes infection in at least 60% of volunteers; safety precludes continuing (>90% AR at 500 CFU) or futility (an AR of 60% is unable to be achieved, even with a 3000 CFU dose). It may take more or less than 3 dose-finding groups to find the optimal dose for which the primary outcome (shigellosis) is achieved in approximately ≥60% of the volunteers and thus the total number of volunteers enrolled in both phases may be less or more than N=60. Once the optimal dose is established in Phase A, that dose will be carried forward for verification in Phase B. For Phase B, dose verification groups of 30 volunteers (2 cohorts of 15 volunteers per cohort) will be conducted to verify the AR with the chosen dose. The dose finding and verification stages will be done in a staggered fashion in case the dose needs to be adjusted, resulting in approximately 5 cohorts to be enrolled over time. Allocation into the groups will be on "first come first served basis" with no randomization occurring for enrolment in any of the cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 45 years of age (inclusive) Kilifi County residents
* Able and willing (in the Investigator's opinion) to comply with all study requirements.
* Provide informed consent.
* Demonstrate comprehension of the protocol procedures and knowledge of study by passing a test of understanding (pass grade 100%).
* Use of effective method of contraception for the entire duration of study (prior to study start and up to study completion) (women only). Female volunteers will be asked to provide their family planning records to verify. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly, in accordance with the product label. Examples of these include: combined oral contraceptives; injectable progestogen; implants of etenogestrel or levonorgestrel; intrauterine device or intrauterine system; male partner sterilisation at least 6 months prior to the female volunteer's entry into the study, and the relationship is monogamous; male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository); and male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository).
* Willingness to participate for an inpatient stay lasting approximately 12 days or longer and an outpatient follow-up lasting about 12 months from challenge.
* Available for all planned follow-up visits.

Exclusion Criteria:

* Presence of a significant medical condition (e.g., psychiatric conditions, alcohol or illicit drug abuse/dependency, or gastrointestinal disease, such as peptic ulcer, symptoms or evidence of active gastritis or gastroesophageal reflux disease, inflammatory bowel disease), or other laboratory abnormalities which in the opinion of the investigator precludes participation in the study.
* Known immunosuppressive illness for example those with cancer, on immunosuppressive therapy, HIV etc.
* Positive serology results for HIV, HBsAg, or HCV antibodies.
* Evidence of inflammatory arthritis on exam and/or HLA-B27 positive.
* Family history of inflammatory arthritis.
* Clinically significant abnormalities in screening lab haematology or serum chemistry, as determined by PI or PI in consultation with the research monitor and Sponsor.
* Known allergies to fluoroquinolones, β-lactams or trimethoprim-sulfamethoxazole (any of the three are exclusionary).
* Fewer than 3 stools per week or more than 3 stools per day as the usual frequency.
* History of diarrhoea in the 2 weeks prior to planned inpatient phase.
* Use of antibiotics during the 7 days before receiving the challenge inoculum dosing.
* Use of prescription and/or OTC medications that contain imodium, acetaminophen, aspirin, ibuprofen, and/or other non-steroidal anti-inflammatory drugs, during the 48 hours prior to investigational product administration.
* Confirmed PCR positive for SARS-COV-2 three days before challenge i.e., Day -3.
* Use of any medication known to affect the immune function within 30 days preceding receipt of the challenge inoculum or planned use during the active study period.
* Serologic evidence of prior S. sonnei infection as determined by ELISA.
* A chronic disease for which doses of prescription medications are not stable for at least the past 3 months.
* Have known immunocompromised household contacts for example those with cancer, on immunosuppressive therapy, HIV etc.
* A clinically significant abnormality on physical examination, including a systolic blood pressure >140 mm Hg or diastolic blood pressure >90 mm Hg, or a resting pulse >100 beats/min or <55 beats/min (<50 beats/min for conditioned athletes).
* Pregnant, nursing, or planning to become pregnant within 29 days of receipt of the study product.
* In the 4 weeks following challenge, volunteer will be living with or having daily contact with elderly persons aged 70 years or more, diapered individuals, persons with disabilities, children <2 years old, a woman known to be pregnant or nursing, or anyone with diminished immunity. This includes contact at work, home, school, day-care, nursing homes, or similar places.
* Work in a health care setting, day care center, or as a food handler in the 4 weeks following the challenge with S. sonnei.
* Use of any investigational drug or any investigational vaccine within 60 days preceding challenge, or planned use during the 6 months after receipt of the study agent.
* Have received a licensed, live vaccine within 28 days or a licensed inactivated vaccine within 14 days of receiving the challenge inoculum.
* Inability to comply with inpatient rules and regulations.
* Has any other condition that, in the opinion of the Investigator, would jeopardize the safety or rights of a volunteer (e.g., infection with another detected pathogen) or would render the volunteer unable to comply with the protocol.
* Received blood or blood products within the past six months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of volunteers with solicited adverse events | Through 11 days post challenge
  Occurrence and severity of solicited adverse events (AEs) through 11 days post-challenge. Occurrence, severity, and relatedness of unsolicited AEs through 11 days post-challenge. Occurrence, severity, and relatedness of serious adverse events (SAEs) throughout the entire study. Occurrence of abnormal clinical laboratory values within 11 days post challenge. Percent of volunteers with nausea, vomiting, anorexia, abdominal pain/cramps rated as moderate to severe.
Number of volunteers with an attack rate of ≥60% | Through 11 days post challenge
  Confirmation of the dose with an acceptable safety profile as determined by that gives an attack rate of ≥60% of shigellosis in Kenyan adults.

SECONDARY OUTCOMES:
Percent of volunteers with | Through 11 days post challenge
  Maximum 24-hour stool output
Percent of volunteers shedding | Through 11 days post challenge
  Peak shedding levels of the 53G challenge strain (CFUs/g of stool) post-challenge based on the results of quantitative cultures post-challenge
Kinetics of serum IgA and IgG antibody responses | From baseline to 366 days
  S. sonnei O-Ag, LPS, IpaB, and IpaC;

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI-Wellcome Trust Research Programme, Kilifi, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Within 2 years of the study completion date
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 2 years of the study completion date